CLINICAL TRIAL: NCT02904967
Title: Identification of New Genetic Markers of Risk of Venous Thromboembolism Recurrence by Analyzing Whole Genome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-30; 2012-A01139-34 (Other: ANSM)
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with recurrent VTE (Experimental)
  Interventions: Biological: Extra Blood Draw
- patients with only one episode of VTE (Active Comparator)
  Interventions: Biological: Extra Blood Draw

INTERVENTIONS:
Biological: Extra Blood Draw

SUMMARY:
Venous thromboembolism (VTE) is a common and potentially fatal disease. It is considered a chronic disease with a recurrence rate of 30% at 10 years.

Reduce the risk of recurrence is a serious public health issue. For this it is necessary to identify patients at high risk of recurrence. However, until now, only 50% of recurrences are in the presence of known risk factors, suggesting that there are still yet unidentified risk factors.

The assumption behind this project is that there are specifically associated genetic polymorphisms to the risk of VTE recurrence.

The aim of our project is to identify these polymorphisms from genome-wide data MARTHA cohort. This cohort is composed of 1542 subjects from the Marseille region with at least one episode of VTE documented. Patients in the cohort MARTHA have all been genotyped for approximately 500,000 polymorphisms.

The investigators want to achieve a case-control study nested in the cohort MARTHA. Subjects with recurrent VTE (the case) will be compared to subjects with only one episode of VTE (the controls). The allelic frequencies of polymorphisms previously genotyped 500,000 will be compared between cases and controls. The identification of these new genetic variants associated with VTE recurrence should allow us to improve the pathophysiological knowledge of the disease, reduce the frequency of episodes and focus research on new therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian topic
* Personal history of VTE confirmed by the reference diagnostic tests

Exclusion Criteria:

* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
allelic frequency of 500,000 already genotyped polymorphisms | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No